CLINICAL TRIAL: NCT03112707
Title: Performance of Bioresorbable Polymer-Coated Everolimus-Eluting Synergy® Stent in Patients at High Bleeding Risk Undergoing Percutaneous Coronary Revascularization Followed by 1-Month Dual Antiplatelet Therapy
Brief Title: Bioresorbable Polymer-Coated EES in Patients at High Bleeding Risk Undergoing PCI Followed by 1-Month DAPT
Acronym: POEM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Humanitas Hospital, Italy (Other)
Responsible Party: Principal Investigator, Giulio Stefanini, Assistant Professor of Cardiology, Humanitas Hospital, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 012017POEM
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): 1023 real world high-bleeding risk (HBR) patients with coronary artery disease (stable as well as acute coronary syndromes) who qualify for percutaneous coronary interventions will be included in the study.
  Interventions: Drug: Aspirin; Drug: P2Y12 inhibitor

INTERVENTIONS:
Drug: Aspirin — After percutaneous coronary intervention with bioresorbable polymer-coated everolimus-eluting Synergy® stent implantation, dual antiplatelet therapy with aspirin 100 mg od and a P2Y12 inhibitor will be continued for a duration of 1 month, after which single antiplatelet therapy with aspirin will be recommended indefinitely. In case of need for oral anticoagulation, patients will receive an oral anticoagulant in addition to a P2Y12 inhibitor without aspirin for 30 days.
Drug: P2Y12 inhibitor — After percutaneous coronary intervention with bioresorbable polymer-coated everolimus-eluting Synergy® stent implantation, dual antiplatelet therapy with aspirin 100 mg od and a P2Y12 inhibitor will be continued for a duration of 1 month, after which single antiplatelet therapy with aspirin will be recommended indefinitely. In case of need for oral anticoagulation, patients will receive an oral anticoagulant in addition to a P2Y12 inhibitor without aspirin for 30 days.

SUMMARY:
Objective: To evaluate the safety of bioresorbable polymer-coated everolimus-eluting Synergy® stent followed by 1-month dual antiplatelet therapy in patients at high-bleeding risk.

Study population: Real world high-bleeding risk (HBR) patients with coronary artery disease (stable as well as acute coronary syndromes) who qualify for percutaneous coronary interventions.

Study size: A total of 1023 patients will be enrolled. Study design: Prospective, single-arm, multicentre trial, powered for non-inferiority with respect to objective performance criteria (OPC).

Antiplatelet therapy: Dual antiplatelet therapy with aspirin 100 mg od and a P2Y12 inhibitor for a duration of 1 month, after which single antiplatelet therapy with aspirin will be recommended indefinitely. In case of need for oral anticoagulation, patients will receive an oral anticoagulant in addition to a P2Y12 inhibitor without aspirin for 30 days.

Primary endpoint: Composite of cardiac death, myocardial infarction, or definite/probable stent thrombosis at 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

All patients will need to have symptomatic coronary artery disease including patients with chronic stable angina, silent ischemia, or acute coronary syndromes (including NSTE-ACS and STE-ACS) and presence of one or more coronary artery stenoses >50% in a native coronary artery or a saphenous bypass graft that treated with one or multiple Synergy® stents.

Moreover, in order to be included patients will need to meet at least 1 of the following HBR criteria:

1. Age ≥75 years
2. Oral anticoagulation planned to continue after PCI
3. Hemoglobin <11 g/l,
4. Transfusion within 4 week before inclusion
5. Platelet count <100'000
6. Hospital admission for bleeding in previous 12 months
7. Stroke in previous 12 months
8. History of intracerebral hemorrhage
9. Severe chronic liver disease
10. Creatinine clearance <40 ml/min
11. Cancer in previous 3 years
12. Planned major surgery in next 12 months
13. Glucocorticoids or NSAID planned for >30 days after PCI
14. Expected non-adherence to >30 days of dual antiplatelet therapy

Exclusion Criteria:

1. Cardiogenic shock
2. Major active bleeding at the time of PCI
3. Expected non-adherence with 1 month DAPT
4. Known intolerance to aspirin, clopidogrel, or ticagrelor
5. Inability to provide informed consent
6. Currently participating in another trial before reaching first endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1023 (Estimated)
Dates: Start 2017-04-14 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | 1 year
  Composite of cardiac death, myocardial infarction, and definite/probable stent thrombosis

SECONDARY OUTCOMES:
All-cause death | 30 days and 1 year
  All-cause death
Cardiac death | 30 days and 1 year
  Cardiac death
Myocardial infarction | 30 days and 1 year
  Myocardial infarction (defined according to III universal definition)
Stent thrombosis | 30 days and 1 year
  Stent thrombosis (defined according to ARC criteria)
Target-vessel revascularization | 30 days and 1 year
  Target-vessel revascularization (any and clinically driven)
Target-lesion revascularization | 30 days and 1 year
  Target-lesion revascularization (any and clinically driven)
Major bleeding | 30 days and 1 year
  Major bleeding (BARC 3 to 5)
Cerebrovascular event | 30 days and 1 year
  Cerebrovascular event
Target-lesion failure | 30 days and 1 year
  composite of cardiac death, target-vessel myocardial infarction, or clinically-driven target-lesion revascularization
Patient oriented composite endpoint | 30 days and 1 year
  Composite of any death, any MI, any revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pivato CA, Mincione G, Gramss L, Pacchioni A, Piccolo R, Musto C, Sardella G, Indolfi C, Antonelli G, Regazzoli D, Paradies V, Reimers B, Condorelli G, Testa L, Briguori C, Stefanini G. Early oral anticoagulation monotherapy after PCI: Insights from the POEM trial. Am Heart J. 2026 Mar;293:107309. doi: 10.1016/j.ahj.2025.107309. Epub 2025 Nov 19. PMID 41271123
- [Derived] Maurina M, Pivato CA, Kunadian V, Testa L, Briguori C, Pacchioni A, Latini AC, Cesani N, Piccolo R, Musto C, Sardella G, Indolfi C, Regazzoli D, Paradies V, Stefanini G. One-month DAPT after biodegradable-polymer everolimus-eluting stent implantation in women at high-bleeding risk: Insights from the POEM trial. Catheter Cardiovasc Interv. 2024 Nov;104(6):1129-1138. doi: 10.1002/ccd.31255. Epub 2024 Oct 3. PMID 39359172
- [Derived] Pivato CA, Reimers B, Testa L, Pacchioni A, Briguori C, Musto C, Esposito G, Piccolo R, Lucisano L, De Luca L, Conrotto F, De Marco A, Franzone A, Presbitero P, Ferrante G, Condorelli G, Paradies V, Sardella G, Indolfi C, Condorelli G, Stefanini GG. One-Month Dual Antiplatelet Therapy After Bioresorbable Polymer Everolimus-Eluting Stents in High Bleeding Risk Patients. J Am Heart Assoc. 2022 Mar 15;11(6):e023454. doi: 10.1161/JAHA.121.023454. Epub 2022 Feb 3. PMID 35114814